CLINICAL TRIAL: NCT00671931
Title: Susceptibility of Motor-Evoked Potentials to Varying Targeted Blood Levels of Dexmedetomidine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 06-09-12
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Scoliosis
Keywords: dexmedetomidine; neuromonitoring; spine procedures; safe dose; 1- safe dose of dexmedetomidine when used in total intravenous anesthesia for procedures require neuromonitoring; 2- safe dose of propofol when uses in comination with dexmedetomidine in neuromontoring; 3effect of dexmedetomidine on somatosensory evoked potential and motor evoked potentials
MeSH Terms: conditions — Scoliosis | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- I (Active Comparator): Dexmedetomidine low infusion, Propofol low infusion
  Interventions: Drug: low dexmedetomidine, low propofol
- II (Active Comparator): Dexmedetomidine high infusion, Propofol low infusion
  Interventions: Drug: high dexmedetomidine, low propofol
- IV (Active Comparator): Dexmedetomidine high infusion, Propofol high infusion
  Interventions: Drug: Dexmedetomidin
- V (Active Comparator): Dexmedetomidine intermediate infusion, Propofol intermediate infusion
  Interventions: Drug: Dexmedetomidine
- III (Active Comparator): Dexmedetomidine low infusion, Propofol high infusion
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: low dexmedetomidine, low propofol — Dexmedetomidine loading dose 0.6 MCG/KG,Propofol infusion 100 MCG/KG/M
  Arms: I
Drug: high dexmedetomidine, low propofol — Dexmedetomidine loading dose 1.1 MCG/KG ,Propofol infusion 100 MCG/KG/M
  Arms: II
Drug: Dexmedetomidine — Dexmedetomidine loading dose 0.6 MCG/KG,Propofol infusion 200 MCG/KG/M
  Arms: III
Drug: Dexmedetomidin — Dexmedetomidine loading dose 1.1 MCG/KG.Propofol infusion 200 MCG/KG/M
  Arms: IV
Drug: Dexmedetomidine — Dexmedetomidine loading dose 0.9 mcg/kg,Propofol infusion 140 mcg/kg/min
  Arms: V

SUMMARY:
Reduction of the spinal cord injuries during scoliosis surgery is a major goal of the anesthesia and surgical team. Despite improvement in scoliosis surgery over the years, the development of neurological deficits remains the most feared complication of spine surgery. During scoliosis surgery it is very important to monitor the spinal cord to detect spinal cord injury with surgical manipulation. Continuous or intermittent intraoperative electrophysiological monitoring (neuron-monitoring) is used routinely during these procedures to provide the surgeon with information concerning the integrity of neurological structures at risk. All neuron-monitoring modalities are affected by the anesthetic regimen used. Of the various intravenous anesthetic drugs, the combination of propofol, remifentanil and dexmedetomidine appear to impact neuron-monitoring the least. The current anesthetic practice is to use the three drugs in combination at doses that do not depress the signals but there is no data relating targeted dexmedetomidine and propofol blood levels to neuron-monitoring signals. The lack of data results in wide variability in dosing with consequent variability in patient response.

Hypothesis: Clinically relevant blood levels of dexmedetomidine will affect the amplitude of transcranial motor-evoked potentials (TcMEP) either independently or by interaction with propofol in a dose dependent manner.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 10 to 25 years of age
* Diagnosis of idiopathic scoliosis is established
* Subject's legal authorized representative has given written, informed consent to participate in the study and, where appropriate, the subject has given assent to participate
* American society of Anesthesiology physical status one/two
* Patients scheduled for posterior spinal fusion only

Exclusion Criteria:

* • Patients with neuromuscular scoliosis and patients with motor or sensory deficit in the lower extremities

  * Patients with allergy to, or contraindication for the drugs or techniques used in the study
  * Morbid obesity (Body mass index higher than 40)
  * History of malignant hyperthermia
  * Patient with severe cardiopulmonary disease (pulmonary hypertension, cardiomyopathy, mechanical ventilation)

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahmoud, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinati Children Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Mahmoud M, Sadhasivam S, Salisbury S, Nick TG, Schnell B, Sestokas AK, Wiggins C, Samuels P, Kabalin T, McAuliffe J. Susceptibility of transcranial electric motor-evoked potentials to varying targeted blood levels of dexmedetomidine during spine surgery. Anesthesiology. 2010 Jun;112(6):1364-73. doi: 10.1097/ALN.0b013e3181d74f55. PMID 20460997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment has been completed for this study.
Pre-assignment Details: There is no wash out, run-in, or transition period in this protocol
Groups:
- Low Dexmedetomidine/Low Propofol; High Dexmedetomidine/Low Propofol; Low Dexmedetomidine/High Propofol; High Dexmedetomidine/High Propofol; Intermediate Dexmedetomidine/Intermediate Propofol: Dexmedetomidine Loading Dose, Propofol Loading Dose and Data Collection: After baseline TcMEP measurements are obtained, subject will receive their assigned dexmedetomidine loading dose over a 15 minute period. During this time period, if the subject has been randomized to a Propofol loading dose they will be give it over a 3 minutes period. See Table 2.
  TABLE 2: dexmedetomidine and propofol dose schedule.
  Dexmedetomidine loading dose mcg/kg Dexmedetomidine infusion mcg/kg/hour for 15 minutes Target dexmedetomidine concentration ng/ml (** ) Propofol loading dose mg/kg Propofol infusion mcg/kg/min Target propofol concentration mcg/ml Group 1 0.6 0.4 0.4 none 100 2.5 Group 2 1.1 0.7 0.8 none 100 2.5 Group 3 0.6 0.4 0.4 0.5 200 5.0 Group 4 1.1 0.7 0.8 0.5 200 5.0 Group 5 0.9 0.5 0.6 0.25 140 3.75
Period: Overall Study
Arm/Group | Low Dexmedetomidine/Low Propofol | High Dexmedetomidine/Low Propofol | Low Dexmedetomidine/High Propofol | High Dexmedetomidine/High Propofol | Intermediate Dexmedetomidine/Intermediate Propofol
Started | 9 | 8 | 9 | 10 | 8
Completed | 8 (Nueromonitoring equipment falure) | 8 (All completed) | 9 (all completed) | 8 (Prepositioning - Neuromonitoring required) | 7 (Low heart rate requiring treatment)
Not Completed | 1 | 0 | 0 | 2 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dexmedetomidine/Low Propofol | High Dexmedetomidine/Low Propofol | Low Dexmedetomidine/High Propofol | High Dexmedetomidine/High Propofol | Intermediate Dexmedetomidine/Intermediate Propofol | Total
Number analyzed (Participants) | 9 | 8 | 9 | 10 | 8 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 9 | 10 | 8 | 43
  Between 18 and 65 years | 1 | 0 | 0 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 16 (2) | 15 (2) | 15 (2) | 15 (2) | 15 (2) | 15 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 9 | 9 | 7 | 35
  Male | 5 | 2 | 0 | 1 | 1 | 9
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 9 | 10 | 8 | 44

OUTCOME MEASURES:

1. Primary Outcome: Motor Evoked Potential Amplitude
Description: The primary outcome measure of the study was the participants who had Motor Evoked Potentials Amplitude significantly reduced (more than 70%)compared to the baseline.
Time Frame: baseline, 30 minutes
Measure: Number; unit: participants
Arm/Group | Low Dexmedetomidine/Low Propofol | High Dexmedetomidine/Low Propofol | Low Dexmedetomidine/High Propofol | High Dexmedetomidine/High Propofol | Intermediate Dexmedetomidine/Intermediate Propofol
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 7
participants | 1 | 3 | 1 | 4 | 4

ADVERSE EVENTS:
Arm/Group | Low Dexmedetomidine/Low Propofol | High Dexmedetomidine/Low Propofol | Low Dexmedetomidine/High Propofol | High Dexmedetomidine/High Propofol | Intermediate Dexmedetomidine/Intermediate Propofol
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No